CLINICAL TRIAL: NCT01765309
Title: A Randomized Controlled Trial To Evaluate The Use Of Botox In Breast Reconstruction With Tissue Expanders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-0782
Record Dates: First submitted 2013-01-08; First posted 2013-01-10 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2012-03

CONDITIONS: Breast Cancer
Keywords: Tissue expanders; Botulinum toxin; Botox
MeSH Terms: conditions — Breast Neoplasms | interventions — Plastic Surgery Procedures; Botulinum Toxins; Botulinum Toxins, Type A; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bilateral mastectomy with reconstruction (Experimental): The trial was a comparison between each breast in a single patient undergoing bilateral mastectomy with reconstruction
  Interventions: Procedure: Bilateral mastectomy with reconstruction

INTERVENTIONS:
Procedure: Bilateral mastectomy with reconstruction — In each patient enrolled in the study, botulinum toxin was injected into one pectoralis muscle while saline placebo was injected on the opposite side in a randomized blinded fashion
  Other Names: Botulinum toxin (botox) injection

SUMMARY:
Investigation of whether injection of the pectoralis muscle with 100 units botulinum toxin during breast reconstruction with tissue expanders results in decreased pain using a blinded, randomized, controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral mastectomy with immediate tissue expander reconstruction

Exclusion Criteria:

* Unwilling to receive study injections

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Difference between preoperative and postoperative pain scale | 12 weeks
  Patients reported pain in each breast on a visual analog scale of 1-10 at each clinic visit

CONTACTS AND LOCATIONS:
Overall Officials: Joyce K Aycock, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States